CLINICAL TRIAL: NCT04197180
Title: HybridAPC for the Treatment of Gastric Low Grade Intraepithelial Neoplasia (LGIN): a Prospective, Multi-center Study
Brief Title: Hybrid APC for Gastric Low Grade Intraepithelial Neoplasia
Acronym: HybridAPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Shenzhen Hospital of Southern Medical University (Other); The Fifth Affiliated Hospital of Zunyi Medical College (Other)
Responsible Party: Principal Investigator, Philip Wai Yan CHIU, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC 2019.490-T
Record Dates: First submitted 2019-12-11; First posted 2019-12-12 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Gastric Low Grade Intraepithelial Neoplasia
Keywords: Gastric low grade intraepithelial neoplasia; Hybrid APC; Endoscopic Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid Argon Plasma Coagulation (Experimental): The Hybrid-Argon Plasma Coagulation probe combines waterjet technology with Argon Plasma Coagulation. The probe comprises a central water channel for the submucosa injection function and a peripheral gas channel for the Argon Plasma Coagulation function
  Interventions: Procedure: Hybrid Argon Plasma Coagulation

INTERVENTIONS:
Procedure: Hybrid Argon Plasma Coagulation — Argon Plasma Coagulation after water injection for local ablation

SUMMARY:
This cohort study aims to investigate the clinical efficacy and safety of Hybrid APC for treatment of gastric low grade intramucosal neoplasia.

DETAILED DESCRIPTION:
This cohort study aims to investigate the clinical efficacy and safety of Hybrid APC for treatment of gastric low grade intramucosal neoplasia. Successful ablation is defined as no evidence of local recurrence at 12 months after HybridAPC upon follow up endoscopy. This is defined as absence of LGIN, HGIN and cancer in biopsies obtained at all locations during followup endoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Low grade intraepithelial neoplasia of stomach with size≤20 mm
2. Endoscopic diagnosis suspected gastric LGIN with biopsy confirmed gastric LGIN
3. Endoscopic appearance according to Paris classification of Type 0-IIa, IIb or IIc
4. Patients with informed consent

Exclusion Criteria:

1. Patients who had previous endoscopic treatment (including APC, EMR, ESD) for gastric LGIN, HGIN or gastric carcinoma.
2. Endoscopic evidence of ulcer
3. Biopsy confirmed HGIN
4. Endoscopic diagnosis suspected HGIN while biopsy confirmed LGIN
5. Pregnancy
6. informed consent not available

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete ablation of gastric low grade intraepithelial neoplasia | 12 months
  Successful ablation is defined as no evidence of local recurrence at 12 months after HybridAPC upon follow up endoscopy. This is defined as absence of LGIN, HGIN and cancer in biopsies obtained at all locations during followup endoscopy.

SECONDARY OUTCOMES:
Operative time | 1 day
  Time to complete the procedure
Intraoperative bleeding | 1 day
  Bleeding during the procedure as defined by Grade Definition 0 No bleeding
  1. Less bleeding, could be auto-stopped or used by HibridAPC
  2. Stop bleeding by using hot forceps
  3. Stop bleeding by using clips
Pain after procedure | 3 days
  Pain after the procedure as defined by pain score Grade Definition 0 No pain, I Slight pain, II Moderate pain, III Severe pain, IV Extreme pain. V Unbearable pain
Development of new neoplasia | 12, 24 and 36 months
  Development of new neoplasia including low grade intraepithelial neoplasia, high grade intraepithelial neoplasia and advanced gastric cancers
Progression of Low grade intraepithelial neoplasia | 12, 24 and 36 months
  Progression of the development of low grade intraepithelial neoplasia to high grade intraepithelial neoplasia or advanced gastric cancer
Postoperative complications | 7 days
  Development of postoperative complications including bleeding and perforation
Number of HybridAPC procedures required for treatment | 12 months
  The number of Hybrid Argon Plasma Coagulation performed for complete ablation

CONTACTS AND LOCATIONS:
Overall Officials: Philip WY Chiu, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Combined Endoscopy Center, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided